CLINICAL TRIAL: NCT07031362
Title: Effects of Pulmonary Rehabilitation on Distance-Saturation Product and Clinical Outcomes in IPF Patients With and Without Exercise-Induced Desaturation
Brief Title: The Effectiveness of Pulmonary Rehabilitation on Saturation in Patients With Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ilknur Naz, Prof. Dr., Izmir Katip Celebi University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KKK333
Record Dates: First submitted 2025-06-03; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: IPF; Pulmonary Fibrosis
Keywords: fibrosis; pulmonary rehabilitation; exercise training; saturation
MeSH Terms: conditions — Pulmonary Fibrosis; Fibrosis | interventions — Exercise; Dosage Forms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Desaturated Patients (Active Comparator): Patients whose oxygen saturation dropped to 88% or below during the pre-rehabilitation 6MWT were classified as the desaturation group
  Interventions: Other: EXERCISE TRAINING WITH OR WITHOUT MEDICATION
- Non-desaturated group (Active Comparator): Those with oxygen saturation of 89% or above were classified as the non-desaturation group.
  Interventions: Other: EXERCISE TRAINING WITH OR WITHOUT MEDICATION

INTERVENTIONS:
Other: EXERCISE TRAINING WITH OR WITHOUT MEDICATION — All patients who participated in the pulmonary rehabilitation and physiotherapy program underwent sessions lasting approximately two hours, conducted twice weekly over a period of eight weeks. The exercise program included breathing exercises, relaxation and stretching exercises, peripheral muscle strengthening exercises, and aerobic training.

SUMMARY:
The aim of this study is to evaluate the effects of a pulmonary rehabilitation (PR) program on health outcomes and the distance-saturation product in patients with IPF, by comparing two distinct groups: those who experience desaturation and those who do not during the six-minute walk test (6MWT).

DETAILED DESCRIPTION:
Exercise-induced dyspnea and desaturation are distinguishing features of patients with idiopathic pulmonary fibrosis (IPF); these symptoms are associated with disease severity and poorer prognosis. The distance-saturation product, which combines the distance walked and oxygen saturation by multiplying the two measures, has been identified as a predictor of mortality.

Patients with IPF who completed the pulmonary rehabilitation (PR) program were included in the study. Pre- and post-program assessments included spirometric measurements, arterial blood gas values, perception of dyspnea using the Modified Medical Research Council (mMRC) dyspnea scale, exercise capacity via the six-minute walk test (6MWT), health-related quality of life using the St. George's Respiratory Questionnaire (SGRQ) and the Short Form-36 (SF-36), and psychological symptoms assessed with the Hospital Anxiety and Depression Scale (HADS). Additionally, the distance-saturation product was calculated by multiplying the distance walked by the oxygen saturation at the end of the 6MWT. Patients whose oxygen saturation dropped to 88% or below during the pre-rehabilitation 6MWT were classified as the desaturation group, while those with oxygen saturation of 89% or above were classified as the non-desaturation group. The obtained data were compared between these two groups.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Idiopathic Pulmonary Fibrosis Patients who initiated antifibrotic therapy Patients who completed the pulmonary rehabilitation program.

Exclusion Criteria:

* Kardiovascular comorbid conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Exercise capacity | up to 8 weeks
  Six minute walk test

SECONDARY OUTCOMES:
Dyspnea Sensation | Before and after the pulmonary rehabilitation programme (up to 8 weeks)
  Modified Medical Research Council (MMRC)" dyspnea scale, which consists of 5 items ranging between 1 and 5, to determine the severity of patients' shortness of breath. Higher scores mean a worse outcome.
Respiratory Functions | Before and after the pulmonary rehabilitation programme (up to 8 weeks)
  Pulmonary Function Test Pulmonary function test (PFT) which is noninvasive tests that show how well the lungs are working. The tests will measure FEV1; It is the volume of air (in liters) exhaled in the first second during forced exhalation after maximal inspiration.
  FVC: It s the amount of air that can be forcibly exhaled from your lungs after taking the deepest breath possible, as measured by spirometry FEV1/FVC: It represents the proportion of a person's vital capacity that they are able to expire in the first second of forced expiration (FEV1) to the full, forced vital capacity (FVC).
Disease Related Quality of Life Measurement | Before and after the pulmonary rehabilitation programme (up to 8 weeks)
  St. George's Respiratory Questionnaire (SGRQ) to determine disease-specific quality of life. At this scale, high scores define worsened disease and increased symptoms. Higher scores mean a worse outcome.
Health-Related Quality of Life Measurement | Before and after the pulmonary rehabilitation programme (up to 8 weeks)
  Short Form-36 Survey is used to determine health-related quality of life. At this scale, high scores define a better perceived quality of life.
Anxiety and Depression | Before and after the pulmonary rehabilitation programme (up to 8 weeks)
  Hospital Anxiety and Depression Inventory for assessment of anxiety and depression. In this scale; scores of anxiety and depression are calculated separately. The maximum score for both is 21 and high scores correspond to high degree anxiety and depression. Cut-off scores for anxiety and depression were determined as 10/11 and 7/8 respectively.

IPD SHARING:
Plan to Share IPD: No